CLINICAL TRIAL: NCT00345228
Title: Myopic Macular Haemorrhages
Status: Completed | Type: Observational
Sponsor: Singapore National Eye Centre (Other Government)
Other Study IDs: R347/05/2004
Record Dates: First submitted 2006-06-26; First posted 2006-06-27 (Estimated); Last update posted 2006-06-27 (Estimated); Status verified 2004-05

CONDITIONS: Myopic Macular Haemorrhages
Keywords: High myopia; Choroidal neovascularisation; Lacquer crack; Fundus fluorescein angiography; Indocyanine green angiography; Axial length
MeSH Terms: conditions — Choroidal Neovascularization

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
1. To identify the underlying causes of macular haemorrhages in patients with high myopia
2. In the eyes found to have macular haemorrhages secondary to choroidal neovascularisation, we hope to identify the risk factors for the development of choroidal neovascularisation in high myopia
3. To study the functional outcome of these eyes as assessed by visual acuity
4. To study the morphological outcome of these eyes by clinical assessment (and fundal photography) and fluorescein angiography

DETAILED DESCRIPTION:
Primary Aims

* To identify the underlying aetiologies of macular haemorrhages in myopic eyes
* To study the functional and morphological outcome of these eyes with macular haemorrhages 6 months later Secondary Aims
* To study the subgroup of eyes with myopic choroidal neovascularisation (CNV), in particular the risk factors for CNV in myopes
* To study the subgroup of eyes with macular haemorrhages in the absence of CNV

Plan of investigation:

1. Patient with myopia (>-6.00DS) presents with loss of central vision
2. Examination reveals a macular haemorrhage
3. Investigations

   * Refraction
   * Axial length*
   * Fundus fluorescein angiography
   * Indocyanine green angiography*
4. Determine if a myopic CNV is present or absent
5. Management of patient: Treatment vs No treatment

   * Treatment being

     1. Conventional laser
     2. PDT
6. Review at 6 months

   * BCVA
   * Clinical appearance (fundal photo)
   * FFA
7. Review at 12 months

   * BCVA
   * Clinical appearance

ELIGIBILITY:
Inclusion Criteria:

* High myopia (greater than -6.00DS)
* Macular haemorrhage

Exclusion Criteria:

* Macular haemorrhages from other causes eg. diabetic retinopathy, hypertensive retinopathy
* Allergy to fluorescein or indocyanine green dyes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2004-06; Study Completion 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Yen Lee, FRCSEd, Principal Investigator — Singapore National Eye Centre; Chong-Lye Ang, FRCOphth, Study Chair — Singapore National Eye Centre
Locations (1):
- Singapore National Eye Centre, Singapore, Singapore